CLINICAL TRIAL: NCT06111365
Title: A Pivotal, Observational, Prospective Assessment Study to Assess the Performance of Fairtility CHLOE BLAST™ Algorithm for the Prediction of Blastocyst Formation in Women Undergoing In-vitro Fertilization
Brief Title: Pivotal Observational CHLOE Study
Status: Completed | Type: Observational
Sponsor: Fairtility (Industry)
Responsible Party: Sponsor
Other Study IDs: FRT-02-22
Record Dates: First submitted 2023-10-24; First posted 2023-11-01 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: IVF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- IVF: Women undergoing fresh IVF treatment using their own eggs or donor eggs
  Interventions: Device: CHLOE

INTERVENTIONS:
Device: CHLOE — the system will provide to the user a "CHLOE™ score", which is a blastocyst development prediction value, a discrete grading for blastocyst associated with the likelihood of the embryo reaching the blastocyst stage at Day 5

SUMMARY:
This pivotal study is an observational, prospective assessment, multi-center, databank based, clinical study aimed to evaluate the performance of CHLOE™ algorithm in prediction of blastocyst formation.

DETAILED DESCRIPTION:
This pivotal study is an observational, prospective assessment, multi-center, databank based, clinical study aimed to evaluate the performance of CHLOE™ algorithm in prediction of blastocyst formation.

Day 3 morphological grading will be performed by three clinical embryologists (hereafter "Assessors"), who will use standard embryo grading assessment techniques and will be blinded to the CHLOE™ information and to the actual blastocyte status (Yes/No).

Five independent embryologists (hereafter "Panelists") who will be masked to imaging data, to actual blastocyst status, and to each other evaluations will be provided with the morphological grading information performed earlier by the 3 assessors and with the age of subject or egg donor. All data will be presented to Panelists as full cohorts of embryos for each mother. Then they will provide their prediction on blastocyst status of each embryo twice: once the prediction will be based on morphology only and once on morphology plus CHLOE™ assigned score ("High", "Medium+", "Medium-", or "Low"). The two assessments will be done with a washout period of at least 2 weeks and no information will be provided to link the two assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Women undergoing fresh IVF treatment using their own eggs or donor eggs.
2. Women at least 18 years of age; in case of a donor egg the donor shall be at least 18.
3. Total antral follicle count (AFC) of at least 12 as measured by ultrasound prior to stimulation (in cases where AFC is performed).
4. Basal follicle-stimulating hormone (FSH) level < 10 IU or AMH > 1.2 ng/ml
5. At least 8 normally fertilized eggs at bipronuclear (2PN) stage in this in-vitro fertilization cycle.
6. Fertilization using only ejaculated sperm (fresh or frozen) - no surgically removed sperm.
7. At least 2 cells embryo.
8. Embryos were cultured in a Embryoscope ES-D (i.e., EmbryoScope model D - 6 spaces for patients, 12 wells each, resolution - 500*500). The EmbryoScope was configured to the default values provided by EmbryoScope manufacturer.

Exclusion Criteria:

1. Gestational carriers
2. Concurrent participation in another clinical study
3. Previous enrollment in this clinical study (i.e., previous cycles of the same women)
4. History of cancer
5. Use of re-inseminated eggs
6. Embryos that underwent day 3 biopsy for preimplantation genetic testing (PGT)
7. Embryos that underwent biopsy at cleavage stage
8. Non-2PN embryos
9. Embryos with video frames in which the embryo is not clearly visible. Namely, videos with empty well, Bad Focus, Cropped Embryo, Air Bubble (see Annotation protocol, embryos with "Technical Errors" states)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women undergoing fresh IVF treatment using their own eggs or donor eggs
Study Population: Women undergoing fresh IVF treatment using their own eggs or donor eggs
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
The Odds Ratio (OR) for the adjunct prediction of blastulation is required to be statistically significantly greater than 1 | day 5
  The prediction of blastocyst outcome using CHLOE algorithm, and the actual blastocyst outcome for a subset of good/fair embryos will be measured using odds ratio.

SECONDARY OUTCOMES:
The Odds Ratio (OR) for predicting blastocyst formation based on adjunct prediction with CHLOE for all embryos | Day 5
The Odds Ratio (OR) for predicting blastocyst formation using traditional morphology only | Day 5
The Odds Ratio (OR) for Good/Fair embryos predicting blastocyst formation for each individual embryologist | Day 5
Embryo level diagnostic performance measures (Specificity, Sensitivity, Negative predictive value (NPV), Positive predictive value (PPV), Negative likelihood ratio, Positive likelihood ratio) | Day 5

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Weill Cornell Medicine, New York, New York
  - Cleveland Clinic Fertility, Cleveland, Ohio
  - Dallas Fertility Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No